CLINICAL TRIAL: NCT06321601
Title: A Phase 3, Open-label, Uncontrolled Single-arm Study to Evaluate the Efficacy, Pharmacokinetics, and Safety of Avacopan in Combination With a Rituximab or a Cyclophosphamide-containing Regimen in Children From 6 Years to < 18 Years of Age With Active ANCA-associated Vasculitis (AAV)
Brief Title: Study to Evaluate Avacopan in Combination With a Rituximab or Cyclophosphamide-containing Regimen, in Children From 6 Years to < 18 Years of Age With AAV.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230070
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Vasculitis
Keywords: Pediatric; Avacopan; Tavneos®
MeSH Terms: conditions — Vasculitis | interventions — avacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avacopan (Experimental): Participants will receive avacopan twice-daily (BID) administered as oral tablets or liquid formula for 52 weeks.
  Interventions: Drug: Avacopan

INTERVENTIONS:
Drug: Avacopan — Oral administration
  Other Names: AMG 569

SUMMARY:
The main objective of this study is to explore the efficacy of avacopan in participants affected by AAV.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children and adolescents from 6 to < 18 years of age
* Clinical diagnosis of granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA), consistent with Chapel-Hill Consensus Conference definitions (Jennette et al, 2013)
* Newly diagnosed or relapsed AAV with positive test for anti-PR3 or anti-MPO antibodies
* At least 1 PVAS major item, at least 3 PVAS nonmajor items, or at least the 2 renal items of proteinuria and hematuria.
* eGFR > 15 mL/min/1.73 m2 (using modified Schwartz equation per central lab guidelines)
* Participants must have a bodyweight of ≥ 15 kg at day 1.

Exclusion Criteria:

* Any other known multisystem autoimmune disease including eosinophilic granulomatosis with polyangiitis (Churg-Strauss), systemic lupus erythematosus , IgA vasculitis (Henoch-Schönlein), rheumatoid vasculitis, Sjogren's syndrome, anti-glomerular basement membrane disease, or cryoglobulinemic vasculitis
* Alveolar hemorrhage requiring invasive pulmonary ventilation support anticipated to last beyond the screening period of the study
* Any medical condition requiring or expected to require continued use of immunosuppressive treatments, including corticosteroids that may cause confoundment with study assessments and study conclusions.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2028-09-26 (Estimated); Study Completion 2028-09-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Disease Remission at Week 26 According to the Pediatric Vasculitis Activities Score (PVAS) | Week 26
Proportion of Participants With Sustained Disease Remission at Week 52 According to the PVAS | Week 52

SECONDARY OUTCOMES:
Plasma Concentrations of Avacopan | Day 1 up to Week 52
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAE) | Day 1 up to approximately Week 60
  TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs. A serious TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s) that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Proportion of Participants Achieving Disease Remission at Week 26 According to the Birmingham Vasculitis Activity Score (BVAS) | Week 26
Proportion of Participants Achieving Disease Remission at Week 52 According to the BVAS | Week 52
Proportion of Participants With PVAS of 0 Over Time Through Week 52 | Up to Week 52
Proportion of Participants With BVAS of 0 Over Time Through Week 52 | Up to Week 52
Change From Baseline Over 52 Weeks in Urinary Albumin-Creatinine Ratio (UACR) | Baseline up to Week 52
Change From Baseline Over 52 Weeks in Estimated Glomerular Filtration Rate (eGFR) | Baseline up to Week 52
Change From Baseline Over 52 Weeks In Physician Global Assessment (PGA) of Disease Activity | Baseline up to Week 52
Change From Baseline Over 52 Weeks in Pediatric Vasculitis Damage Index (PVDI) | Baseline up to Week 52
Number of Glucocorticoid Dosages Administered | Screening up to Week 52
Proportion of Participants Across the Taste Score Categories of the TASTY Faces Scale | Day 1 and Week 2
  The TASTY faces scale will be utilized to assess the taste of the oral pediatric formulation. A 7-point version of the scale will be used, where higher scores correspond to faces showing favorable tastes. Upon drug administration, the child will be shown the TASTY scale and asked to rate his/her perception of tastiness by pointing to the appropriate face on the scale.
Taste and Acceptability Score of Avacopan per TASTY Faces Scale | Day 1 and Week 2
  The TASTY faces scale will be utilized to assess the taste of the oral pediatric formulation. A 7-point version of the scale will be used, where higher scores correspond to faces showing favorable tastes. Upon drug administration, the child will be shown the TASTY scale and asked to rate his/her perception of tastiness by pointing to the appropriate face on the scale.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (10):
  - Emory University, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Minnesota Masonic Childrens Hospital Discovery Clinic, Minneapolis, Minnesota
  - Cohen Children Medical Center, Lake Success, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Charlotte, North Carolina
  - Akron Childrens Hospital, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Upmc Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Childrens Hospital, Houston, Texas
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Gasthuisberg, Leuven
- Canada (3):
  - Alberta Childrens Hospital, Calgary, Alberta
  - Stollery Childrens Hospital, Edmonton, Alberta
  - CHU Sainte Justine, Montreal, Quebec
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Pellegrin, Bordeaux
  - Hospices Civils de Lyon Hopital Femme Mere Enfant, Bron
  - Hopital Necker Enfants Malades, Paris
  - Hopital Necker, Paris
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Dzieciecy Szpital Kliniczny im. Jozefa Polikarpa Brudzinskiego w Warszawie, Warsaw
- Narodny ustav detskych chorob, Bratislava, Slovakia
- Spain (3):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of reevaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com